CLINICAL TRIAL: NCT03700216
Title: Construction of the Evaluation System of Limb Blood Circulation After Fracture of Limbs in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-18-014
Record Dates: First submitted 2018-09-26; First posted 2018-10-09 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Blood Circulation Disorder
Keywords: limb Fracture; limb blood circulation; early-warning model; Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is aimed to construct a multi-parameter early-warning model based on usage of mannitol, using multi-factor regression and combining with previous clinical experience, literature, expert opinions. The investigators will evaluate the predictive value of the model for mannitol usage and gypsum cutting open through cohort study verification.

DETAILED DESCRIPTION:
The investigator will retrospect the data of operative patients with limb fracture in Pediatric Orthopedics Unit of Shanghai Xinhua Hospital in 2016 to collect the basic information about this kind of patient, including age, gender, kind of fracture, temperature and color of skin, swell, artery pulse, laboratory test indicators, method of fixation, and the usage of mannitol. Then, combining the professionals' suggestions, the investigator will use multi-factor regression to identify the independent risk factors of blood circulation disorder. According to the independent risk factors, the early-warning model of blood circulation disorder will be built, and the rating scale as well. Finally, the critical value of blood circulation disorder after limb fracture will be set by receiver operating characteristic curve.

ELIGIBILITY:
Inclusion Criteria:

* Age from 0 to 14 years;
* Children with limb fractures diagnosed by X-ray film;
* The surgical method is open reduction and wire-pin fixation or steel plate internal fixation;
* Children with postoperative plaster fixation;
* Children whose guardian signed informed written consent.

Exclusion Criteria:

* Children with nerve damage which have caused dysfunction such as sensory and motor;
* Children with fracture in other parts or organic diseases.

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with limb fractures diagnosed by X-ray film
Sampling Method: Probability Sample
Enrollment: 201 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Limb Blood circulation disorder | Within 1 year after mannitol treatment
  Number of participants with circulatory disorders (using mannitol treatment) after limb fracture

SECONDARY OUTCOMES:
Number of adverse events | Within 1 year after mannitol treatment
  The adverse events include acute ischemic necrosis, osteofascial compartment syndrome and disability.
Blood oxygen saturation at the end of extremities | Within 1 year after mannitol treatment
  Oxygen saturation is the fraction of oxygen-saturated hemoglobin relative to total hemoglobin (unsaturated + saturated) in the blood, which can reflect the status of blood circulation. Blood oxygen saturation can be get by using percutaneous oxygen saturation monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Ting Zhu, PhD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China